CLINICAL TRIAL: NCT00148447
Title: Placebo-Controlled Trial of Cipralex in the Treatment of Negative Symptoms in Schizophrenia
Brief Title: The Efficacy of Escitalopram for Negative Symptoms in Schizophrenia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: BeerYaakov Mental Health Center (Other Government)
Collaborators: Lundbeck Israel (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Escitalopram-118CTIL
Record Dates: First submitted 2005-09-06; First posted 2005-09-08 (Estimated); Last update posted 2007-05-03 (Estimated); Status verified 2007-02

CONDITIONS: Schizophrenia
Keywords: negative symptoms; depression; ssri; schizophrenia
MeSH Terms: conditions — Schizophrenia; Depression | interventions — Escitalopram

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: escitalopram

SUMMARY:
The aim of this study is to evaluate the therapeutic effect of escitalopram in the treatment of negative symptoms in schizophrenia patients in a double-blind placebo-controlled study.

DETAILED DESCRIPTION:
The aim of this study is to evaluate the therapeutic effect of escitalopram (cipralex) in the treatment of negative symptoms in schizophrenic patients receiving either typical or the newer atypical antipsychotics (olanzapine and risperidone) in a double-blind placebo-controlled study. As there is no drug treatment that is considered as first-line treatment in the treatment of negative symptoms, we thought that the comparison with placebo is plausible. However, it is important to note that the patients will receive the commonly used treatment for their disorder (i.e. antipsychotic medication).

ELIGIBILITY:
Inclusion Criteria:

* Chronic schizophrenia patients,
* Age <60,
* Medicated,
* Inpatients and outpatients,on stable doses of antipsychotic medications for at least one month before the study entry.
* Patients will be clinically stable and free of any additional axis I diagnosis or significant medical illnesses before enrollment into the study.
* A Positive and Negative Syndrome Scale (PANSS) score of 50 or above will be required for entry to the study.

Exclusion Criteria:

* Comorbidity with mania or major depression,
* Pregnancy,
* Lactation,
* Impaired renal or hepatic function,
* History of sensitivity to cipramil or to other drugs from the selective serotonin reuptake inhibitor (SSRI) group.
* Additional exclusion criteria will consist of mental retardation, organic conditions (brain tumors, drug abuse) and severe exacerbation of the psychiatric condition (i.e. suicide attempt, severe psychotic exacerbation) as defined by hospitalization in high-security units, clinical impression and CGI scores of "condition much worsened".
* Patients will be excluded during the study if they will remove their informed consent.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40
Dates: Start 2004-11; Study Completion 2005-09

PRIMARY OUTCOMES:
negative symptoms
social function

SECONDARY OUTCOMES:
positive symptoms
Clinical Global Impression (CGI)
depression

CONTACTS AND LOCATIONS:
Overall Officials: Iulian Iancu, M.D., Principal Investigator — Beer Yaakov Mental Health Center; Moshe Kotler, M.D., Study Chair — Beer Yaakov Mental Health Center
Locations (1):
- Iulian Iancu, Beer Yaakov, Israel

REFERENCES:
- [Background] Friedman JI, Ocampo R, Elbaz Z, Parrella M, White L, Bowler S, Davis KL, Harvey PD. The effect of citalopram adjunctive treatment added to atypical antipsychotic medications for cognitive performance in patients with schizophrenia. J Clin Psychopharmacol. 2005 Jun;25(3):237-42. doi: 10.1097/01.jcp.0000161499.58266.51. PMID 15876902